CLINICAL TRIAL: NCT00896467
Title: Psychological and Emotional Impacts of Participation in Randomized Clinical Studies in Medical Oncology
Brief Title: Psychological and Emotional Impact in Patients Undergoing Treatment For Metastatic Cancer Either in a Clinical Trial or as Standard Off-Trial Therapy
Status: Terminated | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: COL-0701; CDR0000626737 (Registry Identifier: PDQ (Physician Data Query)); COL-IPSY; COL-RCB 2007-A00223-50; INCA-RECF0480
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Anal Cancer; Anxiety Disorder; Breast Cancer; Depression; Esophageal Cancer; Gallbladder Cancer; Gastric Cancer; Kidney Cancer; Liver Cancer; Lung Cancer; Pancreatic Cancer; Small Intestine Cancer
Keywords: anxiety disorder; depression; stage IV breast cancer; stage IV renal cell cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; stage IV gastric cancer; stage IV anal cancer; stage IV pancreatic cancer; stage IV esophageal cancer; advanced adult primary liver cancer; unresectable gallbladder cancer; small intestine cancer
MeSH Terms: conditions — Anus Neoplasms; Anxiety Disorders; Breast Neoplasms; Depression; Esophageal Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Kidney Neoplasms; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Other: questionnaire administration
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information from patients who received treatment for metastatic cancer while participating in a phase II or phase III randomized clinical trial and from patients receiving standard treatment off-trial may help doctors learn more about the psychological and emotional results of being in a clinical trial.

PURPOSE: This clinical trial is comparing the psychological and emotional impact of participating in a randomized clinical trial with the impact of standard treatment in patients with metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the psychological and emotional consequences in patients who underwent first-line antitumor treatment (chemotherapy or targeted therapy) for metastatic disease while participating in a phase II or III randomized clinical trial vs patients who underwent standard first-line treatment off-trial.

Secondary

* To measure and compare the temporal variation of psychological and emotional consequences during and after completion of or stopping of treatment.
* To measure and compare the degree of knowledge of the implications of participating in a clinical study vs the benefits of standard off-trial treatment and evaluate the impact on psychological and emotional experience.
* To evaluate the relationship between the use of adjustment strategies and emotional regulation and psychological and emotional experiences in both of these situations.

OUTLINE: This is a multicenter study.

Patients complete four questionnaires, including assessment of symptoms of anxiety and depression (HADS), quality of life (QLQ-30), adjustment strategies (WCC), and regulation of emotional behavior (ERQ), during their first course of treatment, after the first evaluation of treatment effectiveness, and one week after completion of treatment. During their first evaluation, patients also complete a questionnaire on the modalities of randomized clinical trials and their impact on care (ICEC-R).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer

  * Metastatic disease for which the median progression-free survival is ≥ 4 months
  * Breast, digestive, kidney, lung
* Receiving first-line antitumor therapy (i.e., chemotherapy or targeted therapy) as part of either:

  * Phase II or III randomized clinical trial
  * Standard treatment off-trial

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-3 or Karnofsky PS 50-100%
* No psychological or physical inability to respond to a questionnaire

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No psychotropic treatment, except for antidepressants, anxiolytics, or sleeping pills taken for more than 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Quality of life as assessed by the QLQ-30 questionnaire
Symptoms of anxiety and depression as assessed by the HADS questionnaire
Adjustment strategies and emotional regulation as assessed by the WCC and ERQ questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Clisant — Centre Oscar Lambret
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille
  - Laboratoire URECA, Villeneuve-d'Ascq